CLINICAL TRIAL: NCT01677481
Title: Randomized Evaluation of Vascular Entry Site and Radiation Exposure: REVERE Trial.
Acronym: REVERE
Status: Completed | Type: Observational
Sponsor: Total Cardiovascular Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: MIL/IMRC/RP/TP/10/2010
Record Dates: First submitted 2012-08-23; First posted 2012-09-03 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Exposure to Ionizing Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Femoral: Coronary angiography procedures performed using transfemoral access
- Left radial access: Coronary angiography procedures performed using left radial access site.
- Right radial Access: Coronary angiography procedures performed using Right radial access site.

SUMMARY:
The study compares radiation exposure parameters between coronary angiography procedures performed by left wrist, right wrist or groin (femoral) procedure access site

DETAILED DESCRIPTION:
Patients referred for coronary angiography will be randomized to either left radial, right radial or femoral arterial access sites, and the coronary angiogram will be performed in a standard fashion, including left ventriculography. Radiation exposure parameters including Air Kerma, Dose-area product, Fluoroscopy time and Operator radiation exposure will be recorded. Operator experience as well as demographic data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing diagnostic coronary angiography

Exclusion Criteria:

* non-availability of one or more of the three access sites History of coronary artery bypass graft surgery Need for percutaneous coronary intervention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for diagnostic coronary angiography
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2011-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Air Kerma | 1 day
  The investigators will measure Air Kerma (cumulative) at the end of the procedure of coronary angiography.

OTHER OUTCOMES:
Operator radiation exposure | 1 day
  operator radiation exposure will be measured by a personal dosimeter worn by the operator outside the lead apron on the vest pocket.

CONTACTS AND LOCATIONS:
Overall Officials: Tejas M Patel, MD, DM, Principal Investigator — Chief
Locations (1):
- V.S. General Hospital, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pancholy SB, Joshi P, Shah S, Rao SV, Bertrand OF, Patel TM. Effect of Vascular Access Site Choice on Radiation Exposure During Coronary Angiography: The REVERE Trial (Randomized Evaluation of Vascular Entry Site and Radiation Exposure). JACC Cardiovasc Interv. 2015 Aug 17;8(9):1189-1196. doi: 10.1016/j.jcin.2015.03.026. Epub 2015 Jul 22. PMID 26210808